CLINICAL TRIAL: NCT03837392
Title: A Pilot Study Examining the Efficacy of Brief Acceptance and Commitment Therapy (ACT) for Perinatal Anxiety
Brief Title: Efficacy of Brief Acceptance and Commitment Therapy (ACT) for Perinatal Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Iowa (Other)
Responsible Party: Principal Investigator, Emily Thomas, Clinical Assistant Professor, University of Iowa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 202002658
Record Dates: First submitted 2019-02-08; First posted 2019-02-12 (Actual); Last update posted 2023-07-12 (Actual); Status verified 2023-07

CONDITIONS: Post Partum Depression; Perinatal Depression; Post Partum Anxiety; Perinatal Anxiety
Keywords: Pregnancy; Mental Health
MeSH Terms: conditions — Depression, Postpartum; Psychological Well-Being | interventions — Gravidity; Postpartum Period

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acceptance and Commitment Therapy (Experimental): Acceptance and Commitment Therapy (ACT) - participants in this arm will take part in an online ACT + psychoeducation intervention. The intervention will provide psychoeducation surrounding perinatal anxiety and depression as well as on engaging social support and coping strategies. The ACT portion of the intervention will focus on developing psychological flexibility, which is defined as behaviorally pursuing one's values even in the presence of barriers (e.g., thoughts, emotions). Following the online intervention, the participants will be contacted for two phone coaching calls -- each lasting about 30-45 minutes.
  Interventions: Diagnostic Test: Baseline Assessment (18-26 weeks pregnant); Behavioral: Online Intervention and Phone Coaching Interventions; Diagnostic Test: Follow Up Assessments: 34-36 weeks pregnant and 4-week postpartum; Diagnostic Test: Follow Up Assessments: 8 weeks postpartum
- Supportive Psychoeducation (Active Comparator): Control group - participants in this arm will take part in an online psychoeducation and support intervention. This intervention will focus on psychoeducation surrounding perinatal anxiety and depression, as well as on engaging social support and coping strategies. Following the online intervention, the participants will be contacted for two phone coaching calls -- each lasting about 30-45 minutes.
  Interventions: Diagnostic Test: Baseline Assessment (18-26 weeks pregnant); Behavioral: Online Intervention and Phone Coaching Interventions; Diagnostic Test: Follow Up Assessments: 34-36 weeks pregnant and 4-week postpartum; Diagnostic Test: Follow Up Assessments: 8 weeks postpartum

INTERVENTIONS:
Diagnostic Test: Baseline Assessment (18-26 weeks pregnant) — At baseline, participants will complete several interviews and questionnaires online and via phone to determine psychological history, current functioning, history of trauma, coping styles, and demographic variables.
Behavioral: Online Intervention and Phone Coaching Interventions — ACT is a cognitive-behavioral therapy that seeks to promote psychological flexibility. The active comparator is the Supportive Control. Two phone coaching sessions will occur 2- and 4-weeks post-intervention in both conditions.
Diagnostic Test: Follow Up Assessments: 34-36 weeks pregnant and 4-week postpartum — The follow-up assessments at 34-36 weeks pregnancy and 4-weeks postpartum will be completed via REDCap, an online secure survey platform in order to reduce participant burden.
Diagnostic Test: Follow Up Assessments: 8 weeks postpartum — The follow-up assessment at 8-weeks postpartum will be completed via phone.

SUMMARY:
This protocol will test the hypothesis that Acceptance and Commitment Therapy (ACT) is effective in reducing anxiety and depressive symptoms during the perinatal and postpartum periods. Participants should expect their participation in the study to last 9-12 months.

DETAILED DESCRIPTION:
The study's major theme is "to examine the efficacy of a brief Acceptance and Commitment Therapy (ACT) intervention in treating perinatal anxiety symptoms, as compared to a supportive control condition."

The perinatal and postpartum periods are known to be a vulnerable time for the development of mental health symptomatology, with approximately 7% of women developing postpartum depression in the first three months following childbirth. One known predictor of postpartum depression is perinatal anxiety and distress. The impact of postpartum depression extends beyond the mother, whose distress and daily functioning are affected, with adverse effects on infant development and care. The need for interventions and preventive interventions has been widely indicated for over two decades.

This protocol will describe two conditions, the effects of which will be contrasted to determine the efficacy of ACT in treating anxiety and depressive symptoms among perinatal women. The ACT condition will be compared to a supportive psychoeducation intervention. The effects of the intervention will be determined in terms of self-report measures (anxiety and depressive symptoms, flexibility, mindfulness, social satisfaction) and diagnostic interviews (depression, anxiety). The impact of trauma history and psychodiagnostic history will be examined as moderating factors and/or covariates in the examination of the intervention's efficacy.

This protocol will test the hypothesis that ACT is effective in reducing anxiety and depressive symptoms during the perinatal and postpartum periods. Second, the investigators will examine the intergenerational impact of the intervention on the offspring via offspring birth outcomes, as reported in the electronic medical record. Finally, the investigators will explore mediators and moderators of the treatment outcomes. This work will advance the understanding of the impact of brief interventions on perinatal well-being and improve the ability to disseminate empirically supported interventions for pregnant mothers.

ELIGIBILITY:
Inclusion Criteria:

1. Adult women (ages 18-45) who are between 18-26 weeks pregnant
2. Fluency in English
3. Ability to give informed consent and comply with study procedures (including phone and internet access)
4. Elevated GAD-7 score (10+)
5. Women must be receiving prenatal care
6. Singleton pregnancy

Exclusion Criteria:

1. Prisoners
2. Inability to give informed consent and comply with study procedures
3. Past/current mania, past/current psychoses (assessed with Psychosis Screening Questionnaire)
4. No therapy appointments in last 60 days (not currently in psychotherapy).

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Change in Inventory of Mood and Anxiety Symptoms (IMAS-R) scores from Baseline | Past 1 month
  The IMAS-R provides continuous and diagnostic scores on mood, anxiety, and distress symptoms.

SECONDARY OUTCOMES:
Change in Five Facet Mindfulness Questionnaire | up to 12 month
  This assessment is a 39-item measure where the scale is from 1 (never or rarely true) to 5 (very often or always true). FFMQ measures five facets of mindfulness with respect to one's own experience: observing (8 items), describing (8 items), acting with (8 items), non-judging (8 items), and non-reacting (7 items).
Change in Acceptance and Action Questionnaire (AAQ-2) from Baseline | up to 12 month
  AAQ-2 will be used to measure psychological inflexibility, avoidance behavior, and maladaptive coping. This is a 7 item measure with a scale of 1 (never true) to 7 (always true). Lower scores indicate lesser experiential avoidance.

OTHER OUTCOMES:
Differences in Infant Birth Outcomes | After delivery
  Infant birth outcomes will be obtained from medical records

CONTACTS AND LOCATIONS:
Overall Officials: Emily B K Thomas, PhD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No